CLINICAL TRIAL: NCT01743443
Title: Corneal Sensitivity Changes Following Cross-linking for Progressive Lower Stage Keratoconus
Brief Title: Corneal Sensitivity Cross-linking Keratoconus
Acronym: CSK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, Chairman of IOG, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARVO - BN - 2013
Record Dates: First submitted 2012-12-01; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Keratoconus
Keywords: Corneal sensitivity; Cross-linking; Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sensitiviy (Experimental): Using the Cochet-Bonnet esthesiometer central corneal sensitivity was measured preoperatively, after 7 days, and once a month after surgery until recovery of the baseline preoperative level. Normal levels of central corneal sensitivity were considered above 40mm.
  Interventions: Other: Cochet-Bonnet esthesiometer central corneal sensitivity

INTERVENTIONS:
Other: Cochet-Bonnet esthesiometer central corneal sensitivity — Using the Cochet-Bonnet esthesiometer central corneal sensitivity was measured preoperatively, after 7 days, and once a month after surgery until recovery of the baseline preoperative level. Normal levels of central corneal sensitivity were considered above 40mm.

SUMMARY:
To evaluate corneal sensitivity changes following corneal cross-linking (CXL) in patients with progressive lower stage keratoconus.

DETAILED DESCRIPTION:
Thirty eight eyes of 19 patients (11 women, 8 men) were included in a prospective, nonrandomized clinical study. Mean patient age was 22 years (range, 18-26 years). Inclusion criteria were low stage bilateral progressive keratoconus, transparent cornea and thinnest corneal thickness ≥ 440 µm. Using the Cochet-Bonnet esthesiometer central corneal sensitivity was measured preoperatively, after 7 days, and once a month after surgery until recovery of the baseline preoperative level. Normal levels of central corneal sensitivity were considered above 40mm.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written consent and sign a HIPAA form
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* For females capable of becoming pregnant,agreet o have uurine pregnancy testing performed prior to treatment; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the treatment and continue to use the method until 1 month after the last dose of investigational product.
* Having topographic evidence of keratoconus which is graded as lower stage progressive keratoconus
* Presence of central or inferior steepening on the Pentacam map
* Steepest keratometry (Kmax) value greater than or equal to 51.00D
* BSCVA of 80 letters or fewer for keratoconus on ETDRS chart
* Contact lens wearers only: remove contact lenses one week prior to the screening refraction
* Contact lens wearers only: manifest refraction must be stable between two visits that occur at least 7 days apart

Exclusion Criteria:

* Contraindications, sensitivity or known allergy to the use of the test articles(S) or their components
* If female, be pregnant, nursing, or planning a pregnancy or have a positive urine pregnancy test at Visit 2 prior to treatment or during the course of the study
* Eyes classified as either normal,atypical normal,keratoconus suspect or mild keratoconus on the severity grading scheme
* A history of the insertion of INTACS in the eye to be treated
* A history of previous limbal relaxing incision procedure in the eye to be treated
* Corneal pachymetry that is <350 microns at the thinnest point measured by Pentacam in the eye to be treated
* Eyes which are aphakic
* Eyes which are pseudophakic and do not have a UV blocking lens implanted
* Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications.
* A history of delayed epithelial healing in the eye to be treated
* Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests
* Patients with a currnet condition that, in the investigator's opinion,would interfere with or prolong epithelial healing
* Taking Vitamin C (ascorbic acid) supplements within 1 week of the crosslinking treatment
* A history of previous corneal crosslinking treatment in the eye to be treated
* Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Corneal sensitivity | Central corneal sensitivity was measured preoperatively, after 7 days, and once a month after surgery until recovery of the baseline preoperative level. The avarage was 12 weeks
  To evaluate corneal sensitivity changes following corneal cross-linking (CXL) in patients with progressive lower stage keratoconus.

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, MD PhD, Study Chair — Instituto de Olhos de Goiania
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil